CLINICAL TRIAL: NCT04326270
Title: Crossover Comparison of Tidal Volume Delivery During Nasal Intermittent Positive Pressure Ventilation in Preterm Infants: Infant Cannula vs. Nasal Continuous Positive Airway Pressure Prongs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Ashley L. Lynch, Principle Investigator, Arkansas Children's Hospital Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GR037133
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Respiratory Distress Syndrome in Premature Infant
Keywords: nasal intermittent positive pressure ventilation; non-invasive ventilation; nasal continuous positive airway pressure prongs; infant nasal cannula; tidal volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- nCPAP prongs (Active Comparator)
  Interventions: Device: Nasal interface
- Infant cannula (Active Comparator)
  Interventions: Device: Nasal interface

INTERVENTIONS:
Device: Nasal interface — Randomized to initial interface of nCPAP prongs or infant cannula
  Other Names: Neotech RAM infant cannula; Miniflow Nasal CPAP Prongs

SUMMARY:
Crossover bedside clinical study to examine relative tidal volume delivery during nasal intermittent positive pressure ventilation (NIPPV) and directly compare the RAM® infant cannula to a nasal continuous positive airway pressure (nCPAP) delivery system in vivo. The study population will consist of preterm neonates with mild respiratory insufficiency who are receiving NIPPV, non-invasive neurally adjusted ventilatory assist (NIV NAVA), or nCPAP.

DETAILED DESCRIPTION:
Bedside crossover study of neonates with mild respiratory distress receiving NIPPV. Infants serve as their own controls and are randomized to initial interface of either RAM® infant cannula or Miniflow® nCPAP prongs. Infants are instrumented with the following monitoring equipment: Edi orogastric tube to measure electrical activity of the diaphragm, transcutaneous monitor to measure transcutaneous CO2 and O2, pulse oximeter to measure heart rate and oxygen saturation, and respiratory inductance plethysmography (RIP) bands around the chest and abdomen to measure breathing movements and relative Vt (arbitrary units, a.u.). Data are continuously and simultaneously acquired using a data acquisition system. After 10 minutes of stabilization, infants receive 5 minutes of NIPPV on each of a sequence of four commonly used pressure settings (expressed as peak inspiratory pressure / positive end expiratory pressure): 16/5, 16/8, 20/5, 20/8. This sequence is not randomized and is constant between interfaces. Subjects are then placed on the alternate interface, and the sequence is repeated. Events ("breaths") are separated into 3 types: patient effort synchronized with NIPPV breaths (type I), NIPPV breaths without patient effort (type II), and patient effort without NIPPV breaths (type III).

ELIGIBILITY:
Inclusion Criteria:

* Chronologic age less than 28 days
* Gestational age at birth between 24 weeks 0 days to 34 weeks 6 days
* Currently receiving NIPPV, NIV NAVA, or nCPAP

Exclusion Criteria:

* Oxygen requirement greater than 40%
* Peak inspiratory pressure greater than 20 cm H2O
* Major congenital anomalies of the heart or lungs

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Relative tidal volume delivery, breath type I | 1 hour
  Relative tidal volume measured in arbitrary units (AU) via RIP bands during synchronized breaths
Relative tidal volume delivery, breath type II | 1 hour
  Relative tidal volume measured in arbitrary units (AU) via RIP bands during ventilator-driven breaths
Relative tidal volume delivery, breath type III | 1 hour
  Relative tidal volume measured in arbitrary units (AU) via RIP bands during patient-driven breaths

SECONDARY OUTCOMES:
Ventilator pressure delivery | 1 hour
Ventilator flow delivery | 1 hour
Heart rate | 1 hour
Oxygen saturation | 1 hour
Transcutaneous carbon dioxide tension | 1 hour
Transcutaneous oxygen tension | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lynch AL, Matlock DN, Akmyradov C, Weisner MD, Beck J, Sinderby C, Courtney SE. Tidal volume delivery during nasal intermittent positive pressure ventilation: infant cannula vs. nasal continuous positive airway pressure prongs. J Perinatol. 2024 Feb;44(2):244-249. doi: 10.1038/s41372-023-01846-7. Epub 2023 Dec 21. PMID 38129599